CLINICAL TRIAL: NCT01970852
Title: Addressing Hospital Patient Information Needs Using a Personal Health Record Portal
Brief Title: Addressing Hospital Patient Information Needs Using Information Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); National Library of Medicine (NLM) (NIH)
Responsible Party: Principal Investigator, David Vawdrey, Assistant Professor of Clinical Biomedical Informatics, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAF0264; R01HS021816 (AHRQ); T15LM00707 (Other Grant/Funding Number: National Library of Medicine)
Record Dates: First submitted 2013-10-18; First posted 2013-10-28 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Inpatient
Keywords: Inpatient; PHR Portal; Information Technology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard tablet computer (Experimental): Patient will receive tablet computer within 18 hours of admission and will continue to have access to it for the rest of his/her stay. Tablet has typical applications including access to the internet and entertainment.
  Interventions: Other: Standard tablet computer
- Usual Care (No Intervention): Patients will receive usual care and will answer surveys during the usual time-frame specified.
- Enhanced tablet computer (Experimental): Patients will receive a tablet computer within 18 hours of admission. Tablet will give access to a personalized inpatient personal health record portal. Will also provide access to standard tablet applications (e.g. video calling, streaming movies, etc.)
  Interventions: Other: Enhanced tablet computer

INTERVENTIONS:
Other: Standard tablet computer — No special enhancements or links to personal health information.
  Arms: Standard tablet computer
Other: Enhanced tablet computer — Tablet computer with personalized access to data from the patient's electronic health record.
  Arms: Enhanced tablet computer

SUMMARY:
The aim of this study is to evaluate the impact of an inpatient personal health record (PHR) portal intervention within the hospital environment. The intervention hopes to improve patient engagement with their care and to measure patient activation and satisfaction. Additional clinical measure (e.g. number of adverse events that occur during the stay, changes to medication orders, etc.) will also be studied. Characterization of hospital patient and clinician attitudes towards patient engagement will also be formalized.

DETAILED DESCRIPTION:
This study will utilize an enhanced inpatient PHR portal to allow patients to view their care team, documented allergies and medications (home and hospital) as well as electronically document questions and concerns related to their care. These questions and concerns are visible to members of the patients' care teams within our commercial inpatient electronic health record (EHR). We will study the impact of the technology using a randomized trial of 426 cardiology and cardiothoracic surgery patients at Columbia University Medical Center in Upper Manhattan. We hypothesize that the use of the inpatient PHR portal will identify and address patients' information needs, improve patient activation, engagement and satisfaction, and encourage PHR use after hospital discharge. We also hypothesize that information entered by patients into the PHR portal will be useful to clinicians. There is no compensation for participating in this study.

The specific aims of the proposal are to:

Aim 1: Evaluate the impact of an inpatient PHR portal intervention using a randomized controlled trial. The primary outcomes will be patient activation, engagement and satisfaction. We will also determine whether access to the inpatient PHR portal is correlated with greater use of the PHR after hospital discharge.

Aim 2: Characterize information needs of hospital patients and assess clinicians' attitudes toward patient engagement in the hospital setting. We will analyze the questions and comments that patients record within the PHR portal application and assess the salience of patient-entered information to issues of care quality and safety. This aim will expand our previous work in taxonomy development and hazard and near-miss recognition. A survey will be administered to collect clinicians' perceptions of the barriers to and facilitators of system use. EHR documentation will be reviewed to assess whether patient-entered information was acknowledged by clinicians, and whether changes were made to the patient's plan of care as a result.

ELIGIBILITY:
Inclusion Criteria:

* Speaks English or Spanish
* Admitted to unit where study is ongoing

Exclusion Criteria:

* Does not pass Mini-mental status exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change in Patient Activation Measure | Admission to Unit and 3-5 days after
  The PAM assesses the knowledge, skills and confidence essential to managing one's own health and healthcare. It segments consumers into one of four progressively higher activation levels. The PAM score has been used to predict healthcare outcomes including medication adherence, ER utilization and hospitalization.

SECONDARY OUTCOMES:
Patient Satisfaction | 3-5 days after admission to study
  We will measure patient patient satisfaction using a survey instrument along with data obtained from EHR and PHR system logs. The Patient Survey instrument measures information needs, satisfaction, patient engagement, and system usefulness. It is derived from the 26-item Telemedicine Satisfaction and Usefulness Questionnaire (Bakken, 2006)

CONTACTS AND LOCATIONS:
Overall Officials: David Vawdrey, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Background] Vawdrey DK, Wilcox LG, Collins SA, Bakken S, Feiner S, Boyer A, Restaino SW. A tablet computer application for patients to participate in their hospital care. AMIA Annu Symp Proc. 2011;2011:1428-35. Epub 2011 Oct 22. PMID 22195206
- [Derived] Greysen SR, Magan Y, Rosenthal J, Jacolbia R, Auerbach AD, Harrison JD. Patient Recommendations to Improve the Implementation of and Engagement With Portals in Acute Care: Hospital-Based Qualitative Study. J Med Internet Res. 2020 Jan 14;22(1):e13337. doi: 10.2196/13337. PMID 31934868
- [Derived] Masterson Creber RM, Grossman LV, Ryan B, Qian M, Polubriaginof FCG, Restaino S, Bakken S, Hripcsak G, Vawdrey DK. Engaging hospitalized patients with personalized health information: a randomized trial of an inpatient portal. J Am Med Inform Assoc. 2019 Feb 1;26(2):115-123. doi: 10.1093/jamia/ocy146. PMID 30534990